CLINICAL TRIAL: NCT05828888
Title: Role of Clonal Hematopoiesis of Indeterminate Potential in Endothelial Dysfunction Associated With Heart Failure With Preserved Ejection Fraction
Brief Title: CHIP in Endothelial Dysfunction Associated With HEpEF
Acronym: CHiEF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: INSERM - UMR 1219 (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2022/51; 2023-A00319-36 (Other: N° ID-RCB)
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Clonal Hematopoiesis of Indeterminate Potential (CHIP); Cardiovascular events; Heart Failure; Inflammation; Endothelial dysfunction
MeSH Terms: conditions — Heart Failure; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For all the patients included, 1 specific blood sampling will be performed. These will be taken during a blood sampling realized as part of the follow up of their disease.
  Aliquots not used for mutation research will be used to create a leukocyte DNA library (storage at -20°C) and a plasma library (storage at -80°C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at identifying processes that are deregulated in blood cells by Clonal Hematopoiesis of Indeterminate Potential (CHIP) which are involved in the development of heart failure with preserved ejection fraction (HEpEF).

DETAILED DESCRIPTION:
Heart failure is responsible of 70,000 deaths every year in France. Heart failure can be divided into 2 categories depend on whether the ejection fraction is reduced (HFrEF) or preserved (HFpEF). Most of the treatments efficient in HFrEF are unable to prevent decompensating or reduce mortality associated with HFpEF. HFpEF pathophysiology remains poorly understood, which represents an obstacle to their management and to reduce cardiovascular events they are associated with.

Currently, it is admitted that cardiovascular risk factors (CVRF such as aging, female gender, diabetes mellitus, high blood pressure, hypercholesterolemia, obesity) are responsible of a low grade chronic inflammatory state that causes an endothelial dysfunction that contributes to the development of HFpEF.

However, not all patients with these CVRF develop HFpEF. Moreover, the mechanisms linking CVRF to inflammation or alteration of cardiomyocyte function by endothelial dysfunction remain unknown. This suggests that it exists a role for another factor that remains to be identified.

Clonal Hematopoiesis of Indeterminate Potential (CHIP) result from the acquisition in hematopoietic stem cells of mutations associated with hematological malignancies, in the absence of any hematological disease. This situation initially described with a frequency of <5% before 60 years and >20% after 80 years old appears to be more frequent (>40% of people over 65 years). CHIP are mainly associated with the occurrence of cardiovascular events such as atherothrombosis and heart failure, possibly due to the induction of a chronic inflammation. Because CHIP are very frequent in the elderly and because CHIP are associated with inflammation and cardiovascular events, they could represent the missing link in the pathophysiology sequence that leads to the appearance of endothelial dysfunction and HFpEF development.

ELIGIBILITY:
Inclusion Criteria:

* HFpEF group and control group

  * male or female
  * 50 ≤ age ≤ 85 ans
  * Absence of evidence of hematological malignancy (known or obvious by the results of blood counts)
  * Subject registered with a social security scheme
  * Written informed consent obtained
* HFpEF group

  * patients with a diagnosis of HFpEF according to the criteria defined by the European society of cardiology
* Control group

  * patients with a neuro-cardiovascular pathology without any link to coronaropathy nor heart failure

Exclusion Criteria:

* Hematological malignancy (known or obvious on the results of blood counts)
* Chronic inflammatory disease (cancer, vasculitis, rheumatism, hepato-gastro-intestinal diseases)
* Long term anti-inflammatory treatments:

  * Corticoids
  * Nonsteroidal anti-inflammatory drugs
  * Aspirin (> 325 mg per day)
  * Cyclo-oxygenase II inhibitors
* Persons under judicial safeguards, trustee or curatorship
* Person deprived of judicial or administrative freedom
* Person unable to give her consent
* Non-cooperative person
* Exclusion period after another clinical study or participation to another interventional clinical study testing a drug in the 30 days before inclusion

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. The cohort will be composed of 40 patients with HFpEF and 40 patients without.
  2. Properties of peripheral leukocytes will be studied by scRNA-seq of
     * 3 patients with HFpEF and TET2 mutation
     * 3 patients with HFpEF and DNMT3A mutation
     * 2 patients with HFpEF but without CHIP
     * 3 patients with TET2 mutation but without HFpEF
     * 3 patients with DNMT3A mutation but without HFpEF
     * 2 patients without HFpEF nor CHIP
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Presence of clonal hematopoiesis indeterminate potential (CHIP) | Inclusion Visit
  Presence of CHIP defined as the presence of a mutation with an allele frequency greater than 2%.

SECONDARY OUTCOMES:
Diagnosis of heart failure with preserved ejection fraction | Inclusion Visit
  Diagnosis based on the European Society of Cardiology diagnostic sequence
scRNA-seq analysis | 6 months (+/- 3 months)
  Sixteen patients will be selected for scRNA-seq analysis:
  * 3 patients with HFpEF and TET2 mutation
  * 3 patients with HFpEF and DNMT3A mutation
  * 2 patients with HFpEF but without CHIP
  * 3 patients with TET2 mutation but without HFpEF
  * 3 patients with DNMT3A mutation but without HFpEF
  * 2 patients without HFpEF nor CHIP

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MANSIER, PharmD, Principal Investigator — University Hospital, Bordeaux